CLINICAL TRIAL: NCT05943704
Title: The Frequency of Beef Allergy in Children With Cow Milk Allergy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: FMASU MS322/2022
Record Dates: First submitted 2023-07-06; First posted 2023-07-13 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Cow Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Children with cow milk allergy. (Experimental): Beef introduction for children proven to have cow milk protein allergy
  Interventions: Dietary Supplement: beef broth

INTERVENTIONS:
Dietary Supplement: beef broth — It indicates if the child has allergy of Beef or not.

SUMMARY:
This study aims to determine the frequency of allergy to beef meat in children with allergy to cow's milk by serum measurement. Also, the study aims to assess the sensitivity and specificity of beef IgE in relation to gold standardized of elimination challenge test and to assess effect of eating of cooked meat on symptoms of allergy in those proven to have either CMA alone +/- beef allergy (by serology).

DETAILED DESCRIPTION:
Milk has been recognized as a leading cause for food allergy in children. It is recognized that there is cross-reactivity of bovine serum albumin and bovine γ-globulin which are present in both milk and beef. Thus, children with cow's milk allergy may be instructed to avoid beef.

The true prevalence of beef allergy has been studied only in few research. This current study will add a tertiary center experience in relation of beef allergy to cow's milk protein allergy to fill the gap of knowledge regarding this subject especially in Egypt.

Study Procedures:

Cases will be managed according to the protocol of gastroenterology unit and Allergy, Rheumatology and Immunology Unit, and will be subjected to:

Informed consent: will be obtained from all patient's parents or legal guardians.

All included cases will be subjected to the following phases of the study:

Phase Ⅰ: Recruitment

I. Full medical history taking:

Personal history: Name, age, sex, order of birth, residence, and consanguinity. Complaint.

Present history:

1. Gastrointestinal symptoms

   1. Vomiting (yes/no):

      If yes: onset, course, duration, frequency, force, color, relation to meal, relation to posture and need for IV fluid.
   2. Hematemesis (yes/no):

      If yes: onset, course, duration, frequency, color, need for resuscitation and associated melena.
   3. Diarrhea (yes/no):

      If yes: onset, course, duration, frequency, consistency, blood in stool and straining.
   4. Constipation: (yes/no):

      If yes: onset, course, duration, frequency, consistency, blood in stool and straining.
   5. Other symptoms: colics, nausea, distension, dysphagia, and failure to gain weight.
2. Associated systemic manifestations (Allergic manifestations) including:

   1. Skin allergy (eczema, urticaria, napkin dermatitis).
   2. Chest allergy (wheezing, croup).
   3. ENT manifestations (allergic rhinitis).
   4. Anaphylactic shock.
3. Dietary and nutritional history:

   1. Breast Feeding: (yes/no) If Yes exclusive for how long?
   2. Artificial feeding:

      Age of start, type of formula and indication
   3. Weaning:

Time of start, type of food given (each food and time of introduction especially cow's milk and CMPs) and any problems during weaning (gastrointestinal, respiratory, or skin allergies).

Past history: mode of delivery, NICU admission. Medication history: Type of medications, antireflux medications, laxatives, probiotic.

Family history: atopy, other siblings with CMPA.

II. Careful Clinical examination:

Anthropometric measurements: (weight, height, Wt/Ht ratio and occipto-frontal circumference) Signs of allergy: (atopic dermatitis- allergic rhinitis). Abdominal examination: (Distension-tenderness-organomegaly) Perianal inflammation, napkin rash. All patients suspected of having cow milk allergy will be subjected to elimination re-challenge test (Dupont, 2014).

All patients included in the study were instructed initially to avoid meat products as per protocol of Ain Shams University for 4 weeks.

Blood samples for IgE for beef will be withdrawn at time of enrollment.

Phase Ⅱ:

Patients with history of anaphylaxis will be excluded from this phase. During the oral food challenge (OFC) procedure, patients will be monitored and regularly re-examined prior to each dose and at first signs of reaction. Total dose will be divided into six incremental portions, where every next dose will be double of the previous dose as follows: 1, 2, 4, 8 and 16 g. In case of suspected severe reaction, a much smaller dose was decided (Gonzales González et al. 2018). In cases of anaphylaxis, patients will be given intramuscular epinephrine in the lateral aspect of the thigh and the dose will be calculated based on patient's weight. Dose will be prepared prior to the procedure to avoid any delay.

In case of milder skin reaction or any type of reaction as bronchospasm it will be managed by oral steroids, antihistaminic + any symptom treatment based on what the patient develops. Smaller doses will be given to those who have mild or moderate reaction and those who develop will not continue the OFS.

ELIGIBILITY:
Inclusion Criteria:

* Children from seven months to three years old newly diagnosed with cow milk allergy at Gastroenterology Unit and Allergy, Rheumatology and Immunology Unit.

Exclusion Criteria:

* Critically ill children.
* Patients diagnosed as immune deficiency.
* Patients receiving long term steroid therapy or anti-histaminic.
* Patients who had anaphylaxis or severe reactions from milk
* Patients with skin diseases which can mask skin reactions

Ages: 7 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
Children with Positive IgE for beef. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fiocchi A, Restani P, Riva E, Mirri GP, Santini I, Bernardo L, Galli CL. Heat treatment modifies the allergenicity of beef and bovine serum albumin. Allergy. 1998 Aug;53(8):798-802. doi: 10.1111/j.1398-9995.1998.tb03977.x. PMID 9722230
- [Background] Gonzales-Gonzalez VA, Diaz AM, Fernandez K, Rivera MF. Prevalence of food allergens sensitization and food allergies in a group of allergic Honduran children. Allergy Asthma Clin Immunol. 2018 Jun 18;14:23. doi: 10.1186/s13223-018-0245-x. eCollection 2018. PMID 29946340
- [Background] Espin Jaime B, Diaz Martin JJ, Blesa Baviera LC, Claver Monzon A, Hernandez Hernandez A, Garcia Burriel JI, Merida MJG, Pinto Fernandez C, Coronel Rodriguez C, Roman Riechmann E, Ribes Koninckx C. [Non-IgE-mediated cow's milk allergy: Consensus document of the Spanish Society of Paediatric Gastroenterology, Hepatology, and Nutrition (SEGHNP), the Spanish Association of Paediatric Primary Care (AEPAP), the Spanish Society of Extra-hospital Paediatrics and Primary Health Care (SEPEAP), and the Spanish Society of Paediatric ClinicaL Immunology, Allergy, and Asthma (SEICAP)]. An Pediatr (Engl Ed). 2019 Mar;90(3):193.e1-193.e11. doi: 10.1016/j.anpedi.2018.11.007. Epub 2019 Jan 19. Spanish. PMID 30665859
- [Background] Martelli A, De Chiara A, Corvo M, Restani P, Fiocchi A. Beef allergy in children with cow's milk allergy; cow's milk allergy in children with beef allergy. Ann Allergy Asthma Immunol. 2002 Dec;89(6 Suppl 1):38-43. doi: 10.1016/s1081-1206(10)62121-7. PMID 12487203
- [Background] Martorell A, Plaza AM, Bone J, Nevot S, Garcia Ara MC, Echeverria L, Alonso E, Garde J, Vila B, Alvaro M, Tauler E, Hernando V, Fernandez M. Cow's milk protein allergy. A multi-centre study: clinical and epidemiological aspects. Allergol Immunopathol (Madr). 2006 Mar-Apr;34(2):46-53. doi: 10.1157/13086746. PMID 16606545
- [Background] Paschke A, Besler M. Stability of bovine allergens during food processing. Ann Allergy Asthma Immunol. 2002 Dec;89(6 Suppl 1):16-20. doi: 10.1016/s1081-1206(10)62117-5. PMID 12487199
- [Background] Skypala IJ, Venter C, Meyer R, deJong NW, Fox AT, Groetch M, Oude Elberink JN, Sprikkelman A, Diamandi L, Vlieg-Boerstra BJ; Allergy-focussed Diet History Task Force of the European Academy of Allergy and Clinical Immunology. The development of a standardised diet history tool to support the diagnosis of food allergy. Clin Transl Allergy. 2015 Feb 19;5:7. doi: 10.1186/s13601-015-0050-2. eCollection 2015. PMID 25741437
- [Background] Soares-Weiser K, Takwoingi Y, Panesar SS, Muraro A, Werfel T, Hoffmann-Sommergruber K, Roberts G, Halken S, Poulsen L, van Ree R, Vlieg-Boerstra BJ, Sheikh A; EAACI Food Allergy and Anaphylaxis Guidelines Group. The diagnosis of food allergy: a systematic review and meta-analysis. Allergy. 2014 Jan;69(1):76-86. doi: 10.1111/all.12333. Epub 2013 Dec 14. PMID 24329961
- [Background] Venter C, Brown T, Shah N, Walsh J, Fox AT. Diagnosis and management of non-IgE-mediated cow's milk allergy in infancy - a UK primary care practical guide. Clin Transl Allergy. 2013 Jul 8;3(1):23. doi: 10.1186/2045-7022-3-23. PMID 23835522
- [Background] Werfel SJ, Cooke SK, Sampson HA. Clinical reactivity to beef in children allergic to cow's milk. J Allergy Clin Immunol. 1997 Mar;99(3):293-300. doi: 10.1016/s0091-6749(97)70045-9. PMID 9058683